CLINICAL TRIAL: NCT06266052
Title: the Effects of Four Different Flap Designs on Healing Lower Third Molar Surgery
Brief Title: Evaluation of the Effects of Four Different Flap Designs on Tissue Healing in Lower Third Molar Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Zeynep Gumrukcu, Associate Professor, Recep Tayyip Erdogan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019/04
Record Dates: First submitted 2024-01-15; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Soft Tissue Injuries
Keywords: third molar surgery; flap design; fractal analysis; soft tissue healing
MeSH Terms: conditions — Soft Tissue Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): triangular flep design will be use in third molar impacted surgery
  Interventions: Procedure: Triangular Flap
- Group 2 (Experimental): Berwick flep design will be use in third molar impacted surgery
  Interventions: Procedure: Berwick Flap
- Group 3 (Experimental): Saurez flep design will be use in third molar impacted surgery
  Interventions: Procedure: Saurez Flap
- Group 4 (Experimental): Heitz
  Interventions: Procedure: Heitz Flap

INTERVENTIONS:
Procedure: Triangular Flap — Triangular flap is a type of flap that is made in the retromolar region, from the distal of the 2nd molar tooth towards the ramus and up to the distal gingival sulcus of the 2nd molar, and includes a vertical releasing incision added from the distobuccal sulcus of the 2nd molar tooth. The auxiliary vertical incision made in this flap type allows the wound to be closed without tension.
  Arms: Group 1
Procedure: Berwick Flap — Berwick described a type of flap whose base is in the distolingual direction of the second molar tooth, in which the tongue-shaped vestibular wing extends to the buccal part of the mandible. In this modification, the incision line is not over the bone defect created by the extraction.
  Arms: Group 2
Procedure: Saurez Flap — In the modified flap type he used, Suarez combined the crestal incision (marginal incision) from the distobuccal corner of the second molar tooth, following the line where the retromolar area meets the buccal bone, with a releasing incision made at the mesial and distal ends of the incision.
  Arms: Group 3
Procedure: Heitz Flap — Heitz used the incision line extending from the distobuccal corner of the 2nd molar tooth to the buccal face of the 2nd molar tooth and downwards, by rotating it towards the angulus mandible on the buccal bone.
  Arms: Group 4

SUMMARY:
The aim of this study is to prospectively evaluate the effectiveness of 4 different flap types used during mandibular impacted wisdom teeth surgery on postoperative quality of life, soft tissue and hard tissue healing at the end of the 3rd month.

DETAILED DESCRIPTION:
Patients will be randomly included in 4 groups with 4 different incision types planned among the patients who will apply for impacted third molar tooth extraction, and each group will consist of 25 patients. Triangular flap will be applied to the patients in Group 1, Berwick incision will be applied in Group 2, Suarez incision will be applied in Group 3, and Heitz incision will be applied in Group 4.The operation time will be recorded on the form. The operation time will be evaluated as the period from anesthesia to the last suture. The patient will be called for control on the 2nd and 7th days after the operation. During control periods, pain value will be recorded using a VAS scale numbered between 0 and 10. Parameter data such as trismus, edema, halitosis, color of the healing tissue, presence/type of granulation will be recorded on the forms created during the control periods, and the patients' sutures will be removed on the 7th control day, as is done in impacted third molar surgery. Patients will be called for a check-up at the end of 3 months to detect hard tissue healing, and a panoramic radiography will be taken to check hard tissue healing. Using the patient's 3rd month follow-up x-rays, fractal analysis will be performed in the area to evaluate the quality of the newly formed bone in the extracted tooth area.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 18-45
2. Do not have a systemic disease that prevents tissue healing
3. Patients needed impacted third surgery

Exclusion Criteria

1. Pregancy
2. Allergic conditions
3. Diabetes
4. Smokers
5. Patients with low oral hygiene

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-03-20 (Estimated); Study Completion 2024-04-20 (Estimated)

PRIMARY OUTCOMES:
Eudema Amount | postoperative second and 7.th day
  5 separate length measurements will be made on the face using a flexible ruler. (mm)
Pain Level | postoperative second and 7.th day
  Pain values will be determined with vas scales numbered 0-10.
Trismus Level | postoperative second and 7.th day
  the distance between the incisal edges of the lower and upper teeth during maximum mouth opening will be measured in millimeters with a ruler. (mm)
Halitosis Amount | postoperative second and 7.th day
  It will be evaluated as presence/absence of halitosis. 0/1
bone healing condition | preoperative and postoperative 3th month
  With the help of a program, the amount of trabeculae in the bone will be counted by the box counting method and a numerical value will be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: zeynep gümrükçü, Dr, Study Director — PhD DDS
Locations (1):
- RTEU Faculty of Dentistry, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
no sharing permission